CLINICAL TRIAL: NCT07403773
Title: Comparison of the Effects of Personal Versus Hospital-Provided Dolls on Preoperative Anxiety and Postoperative Delirium in Preschool Children
Brief Title: Personal Versus Hospital-Provided Dolls in Preschool Children
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Filiz Kaya, M.D., Ankara City Hospital Bilkent
Other Study IDs: TABED 1-26-2055
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Preoperative Anxiety; Emergence Delirium in Pediatric Anesthesia
Keywords: Preoperative Anxiety; Emergence Delirium; Pediatric Anesthesia
MeSH Terms: conditions — Emergence Delirium | interventions — Hospitals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hospital-Provided Doll Group: Participants in this cohort will consist of preschool children accompanied by a hospital-provided doll during the preoperative period. Preoperative anxiety levels, serum cortisol concentrations, and postoperative emergence delirium will be assessed as part of routine perioperative observation.
  Interventions: Other: Hospital-Provided Doll
- Personal Doll Group: Participants in this cohort will consist of preschool children accompanied by their own personal doll during the preoperative period. Preoperative anxiety levels, serum cortisol concentrations, and postoperative emergence delirium will be evaluated using standardized assessment tools.
  Interventions: Other: Personal Doll
- No Doll (Control) Group: Participants in this cohort will consist of preschool children who will undergo the surgical process without the use of any doll. Preoperative anxiety, serum cortisol levels, and postoperative emergence delirium will be observed and recorded for comparison purposes.
  Interventions: Other: No Doll

INTERVENTIONS:
Other: Hospital-Provided Doll — Participants will be accompanied by a hospital-provided doll during the preoperative period according to routine clinical practice.
  Other Names: Hospital
  Groups: Hospital-Provided Doll Group
Other: Personal Doll — Participants will be accompanied by their own personal doll during the preoperative period based and routine practice.
  Groups: Personal Doll Group
Other: No Doll — Participants will undergo the surgical process without the use of any doll.
  Other Names: Control
  Groups: No Doll (Control) Group

SUMMARY:
The goal of this study is to evaluate the effects of personal versus hospital-provided dolls on preoperative anxiety and postoperative delirium in preschool children aged 3-7 years undergoing elective adenoidectomy and/or tonsillectomy.

The main questions it aims to answer are:

* Is the use of a personal doll or a hospital-provided doll associated with lower preoperative anxiety compared with no doll use?
* Is dolls used associated with a reduced incidence and severity of postoperative emergence delirium?
* Researchers will compare children accompanied by a hospital-provided doll, children accompanied by their personal doll, and children with no doll to assess differences in preoperative anxiety levels, serum cortisol concentrations, and postoperative delirium scores.

Participants will:

* Be observed in one of three exposure groups (hospital-provided doll, personal doll, or no doll)
* Undergo standardized preoperative anxiety assessments at predefined time points
* Have serum cortisol levels measured during routine intravenous cannulation
* Be assessed for postoperative delirium in the recovery unit

DETAILED DESCRIPTION:
This study is designed to evaluate the association between doll use and preoperative anxiety as well as postoperative emergence delirium in preschool children undergoing elective adenoidectomy and/or tonsillectomy. The study population consists of female children aged 3-7 years who meet the eligibility criteria and are scheduled for elective surgery under general anesthesia.

Participants will be observed in one of three exposure groups based on routine perioperative practice and parental preference: children accompanied by a hospital-provided doll, children accompanied by their personal doll, and children with no doll use. No intervention will be assigned by the investigators, and standard perioperative care will be maintained for all participants.

Preoperative anxiety will be assessed at four predefined time points: in the waiting area (T0), immediately before transfer to the operating room (T1), in the operating room corridor (T2), and just before anesthesia induction (T3). Anxiety levels will be evaluated using the modified Yale Preoperative Anxiety Scale (m-YPAS) and the Visual Analog Scale for Anxiety (VAS-A).

As a biochemical marker of stress response, serum cortisol levels will be measured from an additional blood sample obtained during routine intravenous cannulation performed for clinical purposes. No additional invasive procedures will be required for study-related assessments.

Postoperative emergence delirium will be evaluated using the Pediatric Anesthesia Emergence Delirium Scale (PAED) at three points: immediately after extubation (P0), upon admission to the post-anesthesia care unit (P1), and 30 minutes after admission (P2).

The study aims to provide clinical evidence regarding the potential role of non-pharmacological, easily applicable strategies such as doll use in reducing perioperative anxiety and postoperative delirium in pediatric surgical patients.

ELIGIBILITY:
Inclusion Criteria:

* Female children aged 3-7 years
* Scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia
* Able to communicate verbally
* ASA physical status I or II, according to the American Society of Anesthesiologists classification
* Written informed consent obtained from a parent or legal guardian

Exclusion Criteria:

* Presence of psychiatric, neurological, or developmental disorders
* Presence of chronic pain or ongoing medical treatment that may affect anxiety levels
* Refusal to participate despite repeated encouragement by the investigators
* Use of additional anxiety-reducing methods or medications outside the study protocol prior to intervention
* Previous surgical experience

Ages: 3 Years to 7 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: Female pediatric patients aged 3 to 7 years scheduled for elective adenoidectomy and/or tonsillectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Preoperative Anxiety Level | Waiting area (T0), immediately before transfer to the operating room (T1), operating room corridor (T2), and just before anesthesia induction (T3)
  Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety Scale (m-YPAS) and the Visual Analog Scale for Anxiety (VAS-A) during the preoperative period. Preoperative anxiety will be assessed using m-YPAS, (score range 23-100) and VAS-A (score range 0-10), with higher scores indicating increased anxiety severity.

SECONDARY OUTCOMES:
Postoperative Emergence Delirium | Immediately after extubation (P0), upon admission to the post-anesthesia care unit (P1), and 30 minutes after admission (P2)
  Emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium Scale (PAED; total score range 0-20). A score ≥10 will be considered indicative of emergence delirium, with higher scores reflecting greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, ÇANKAYA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data including demographic characteristics, group assignment, preoperative anxiety scores, and postoperative emergence delirium scores will be shared.
Supporting Information: Study Protocol
Time Frame: Beginning after publication of the primary results and continuing indefinitely.
Access Criteria: De-identified individual participant data and the study protocol will be shared with qualified researchers upon reasonable request and approval by the principal investigator.

REFERENCES:
- [Background] Frenette G, Lessard C, Sullivan R. Selected proteins of "prostasome-like particles" from epididymal cauda fluid are transferred to epididymal caput spermatozoa in bull. Biol Reprod. 2002 Jul;67(1):308-13. doi: 10.1095/biolreprod67.1.308. PMID 12080033
- [Background] Johnson H, Cowey A. Transneuronal retrograde degeneration of retinal ganglion cells following restricted lesions of striate cortex in the monkey. Exp Brain Res. 2000 May;132(2):269-75. doi: 10.1007/s002210000384. PMID 10853951
- [Background] Chamberland C, Bransi M, Boivin A, Jacques S, Gagnon J, Tremblay S. The effect of augmented reality on preoperative anxiety in children and adolescents: A randomized controlled trial. Paediatr Anaesth. 2024 Feb;34(2):153-159. doi: 10.1111/pan.14793. Epub 2023 Nov 4. PMID 37925608
- [Background] Bienfait HM, Baas F, Gabreels-Festen AA, Koelman JH, Langerhorst CT, de Visser M. Two amino-acid substitutions in the myelin protein zero gene of a case of Charcot-Marie-Tooth disease associated with light-near dissociation. Neuromuscul Disord. 2002 Mar;12(3):281-5. doi: 10.1016/s0960-8966(01)00281-4. PMID 11801400

DOCUMENTS (1):
  • Study Protocol (2026-01-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT07403773/Prot_000.pdf